CLINICAL TRIAL: NCT06976879
Title: Intra- and Interindividual Moderators of Prefrontal Excitability Investigated Using Simultaneous TMS With Neuroimaging
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Principal Investigator, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20231218001
Record Dates: First submitted 2025-04-15; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Healthy Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy experimental group: A group of healthy adults shall undergo concurrent 5 Hz iTBS/fMRI measurements
- Active control group: A group of healthy adults shall undergo concurrent 2.5 Hz iTBS/fMRI measurements

SUMMARY:
The simultaneous application of brain stimulation and neuroimaging offers significant potential for advancing basic neuroscience research and developing objective diagnostic and prognostic markers for mental disorders. The University Research Facility in Behavioral and Systems Neuroscience (UBSN), in collaboration with Principal Investigator Dr. Georg Kranz, recently acquired a TMS-compatible Magnetic Resonance Imaging (MRI) radio-frequency head coil. This cutting-edge equipment, developed by Dr. Martin Tik's research lab in Vienna, enables detailed mapping of both local and remote neural effects of intermittent theta-burst stimulation (iTBS)-a non-pharmacological treatment with proven efficacy for mental disorders. The upgraded setup addresses limitations of older concurrent TMS-fMRI systems, which struggled with image quality and practical applicability. The new system incorporates a multi-channel receiver array, allowing for high-resolution imaging at a fast rate. In this design, the TMS coil is positioned outside the imaging coil, with stimulation pulses passing through the thin imaging coil to reach the participant's brain and induce targeted neural changes. This advanced system enables the investigation of therapeutic network changes induced by iTBS by capturing acute brain responses during stimulation. Additionally, its sensitivity allows for dose-response assessments at the individual subject level. To leverage these advancements, pilot studies utilizing concurrent rTMS/fMRI are proposed to investigate intra- and interindividual moderators of therapeutic brain stimulation. The iTBS/fMRI study will focus on stimulation-induced hemodynamic changes in key subcortical structures and networks that mediate therapeutic responses to iTBS. Specifically, the study aims to examine changes in central limbic regions, including the subgenual anterior cingulate cortex (sgACC), anterior insula, amygdala, ventromedial prefrontal cortex, and orbitofrontal cortex. By exploring these regions, the mechanisms underlying the therapeutic effects of rTMS can be elucidated, providing a comprehensive understanding of how acute brain responses translate into clinical outcomes. This approach represents a significant step forward in advancing the understanding of iTBS, with the potential to refine and optimize this treatment for mental disorders.

ELIGIBILITY:
Inclusion Criteria:

* consider yourself healthy in general and aged 18-60

Exclusion Criteria:

* current internal illness;
* current or former psychiatric or neurological illness;
* current or former alcohol or substance abuse;
* current or previous use of any psychotropic medication;
* current or previous use of any illicit drug;
* any ferromagnetic metal in your body;
* known or possible pregnancy, including the situation when the first day of a
* female's last menstrual period was more than 28 days ago; or
* any contraindication to TMS as assessed by Rossi et al.'s (2011) screening questionnaire.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
BOLD signals | Before stimulation (3-5 minutes), during stimulation (3-5 minutes), and post-stimulation (up to 15 minutes after iTBS completion) on visit 2 and visit 3
  This repeated-measures study involves two participant groups. Each participant will attend one screening (visit 1) and two experimental visits (visits 2 and 3), with at least a 48-hour washout period between experimental visits. One group will receive active iTBS and the other active control iTBS during both experimental visits. We will assess iTBS-induced BOLD signal changes in the DLPFC and other brain regions (before, during, and after stimulation) and investigate modulation by interpersonal and day-to-day intrapersonal factors.

SECONDARY OUTCOMES:
Age | visit 1
  Participant's age in years.
Gender | visit 1
  Participant's self-reported gender (e.g., male, female).
Caffeine consumption | Before stimulation on visit 2 and visit 3
  Self-reported caffeine consumption (e.g., number of cups of coffee) prior to the experiment
Mood states | Before stimulation on visit 2 and visit 3
  Mood states will be assessed using the International Positive and Negative Affect Schedule - Short Form (I-PANAS-SF).
  Scale Description: The I-PANAS-SF is a self-report questionnaire consisting of two 5-item subscales: Positive Affect (PA) subscale: Score ranges from 5 (minimum) to 25 (maximum). Higher scores indicate a better outcome (i.e., greater positive affect). Negative Affect (NA) subscale: Score ranges from 5 (minimum) to 25 (maximum). Higher scores indicate a worse outcome (i.e., greater negative affect).
Physical activity | Before stimulation on visit 2 and visit 3
  Assessment of self-reported physical activity level over the last 7 days, measured using the International Physical Activity Questionnaire (IPAQ). The IPAQ asks about the frequency (days) and duration (minutes) of walking, moderate-intensity activities, and vigorous-intensity activities.Self-reported physical activity (e.g., went to the gym or engaged in strenuous exercise before the experiment).
Sleep quality | Before stimulation on visit 2 and visit 3
  Assessment of self-reported subjective sleep quality experienced "the previous night," measured using the Groningen Sleep Quality Scale (GSQS). The GSQS is a 15-item questionnaire (typically 14 items scored) where participants respond "yes" or "no" to questions about their sleep.
Time of the experiment | Before stimulation on visit 2 and visit 3
  The time of day when the experiment was conducted (e.g., morning or afternoon)
Working Memory | After stimulation on visit 2 and visit 3
  Working memory performance as measured with 3-back task
Vigilance | After stimulation on visit 2 and visit 3
  Vigilance levels as measured with the Sustained Attention to Response Task (SART)
Attention | After stimulation on visit 2 and visit 3
  Attention levels as measured with Flanker task
Childhood maltreatment | Visit 1
  Assessment of self-reported history and severity of childhood maltreatment using a 33-item version of the Childhood Trauma Questionnaire (CTQ-33). The CTQ retrospectively measures experiences of emotional, physical, and sexual abuse, and emotional and physical neglect during childhood and adolescence.
Family history in first-degree relatives | Visit 1
  Self-reported family history of mental disorders in first-degree relatives
Marital status | Visit 1
  Participant's self-reported marital status (e.g., single, married, divorced, widowed)
Handedness | Visit 1
  Participant's handedness assessed using the Edinburgh Handedness Inventory (EHI). The EHI is a self-report questionnaire measuring preference for hand use in a series of common activities.
Education years | Visit 1
  Total number of years of formal education completed by the participant

CONTACTS AND LOCATIONS:
Overall Officials: Georg S Kranz, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No